CLINICAL TRIAL: NCT06549088
Title: Analysis of Lung Cancer Tissue With Spatial Frequency Domain Imaging
Acronym: ALCATS
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Hari Keshava, Clinical Assistant Professor, University of California, Irvine
Other Study IDs: 2767
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Lung Diseases; Cancer, Lung
MeSH Terms: conditions — Lung Diseases; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Spatial Frequency Domain Imaging — Resected lung tissue will be removed from the surgical field and labeled with sutures per standard of care. The specimen will then be immediately analyzed using two SFDI devices in the operating room using sterile technique. Each specimen will be recorded up to three times to ensure at least one high fidelity recording is captured. The SFDI data will be analyzed and compared to the official pathology report from the electronic medical record.

SUMMARY:
This study investigates if a new imaging device can detect different types of lung tissue using spatial frequency domain imaging (SFDI). Specifically, this study aims to detect lung nodules within normal lung tissue and determine if lung nodules are cancerous. Patients who have confirmed or suspected lung nodules and who are undergoing resection of those nodules will be recruited for the study. Study participants will undergo standard of care lung nodule resection in the operating room, and the resected specimen will be imaged using the SFDI device immediately after removal from the surgical field. The data captured from the SFDI images will then be compared to the pathology findings to identify optical properties of normal and cancerous lung tissue. Because the intervention is conducted on resected biospecimens, this study yields minimal risk to participants.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years old
* Suspected or confirmed lung nodule on diagnostic imaging
* Undergoing lung resection using an open, endoscopic, or robotic approach
* Standard of care orders placed for a pathology assessment of resected lung tissue
* Adults undergoing lung resection for a lung mass

Exclusion Criteria:

* <18 years old
* Pregnant females and incarcerated individuals
* No standard of care orders to obtain a pathology assessment
* RUSH pathology order for resected lung tissue
* Any condition where the principal investigator determines to impact patient safety or quality of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults undergoing surgical resection of a suspected or confirmed lung mass.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Markers of native lung parenchyma | May 7, 2023 to December 31, 2026
  Use SFDI to identify markers of lung nodule vs native lung parenchyma

SECONDARY OUTCOMES:
Cancer identification | May 7, 2023 to December 31, 2026
  Distinguish cancer vs non-cancer in lung nodules with SFDI

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No